CLINICAL TRIAL: NCT00127504
Title: Trial of Rifampin and Azithromycin for Treatment of Endosymbiotic Bacteria (Wolbachia) in Onchocerca Volvulus in Guatemala
Brief Title: Clinical Trial of Rifampin and Azithromycin for the Treatment of River Blindness
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Universidad del Valle, Guatemala (Other); University of Alabama at Birmingham (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDC-NCID-3843
Record Dates: First submitted 2005-08-04; First posted 2005-08-08 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Onchocerciasis
Keywords: Onchocerciasis; Wolbachia; Therapy
MeSH Terms: conditions — Onchocerciasis | interventions — Rifampin; Azithromycin

INTERVENTIONS:
Drug: Rifampin
Drug: Azithromycin

SUMMARY:
The purpose of this study is to determine whether rifampin and/or azithromycin are effective in the treatment of river blindness (onchocerciasis).

DETAILED DESCRIPTION:
Mass treatment with ivermectin (Mectizan, Merck & Co) is the mainstay of the current efforts to control onchocerciasis, but the drug is not lethal to adult Onchocerca volvulus parasites. Wolbachia, an endosymbiotic bacterium necessary for the fecundity of O. volvulus, can be eradicated with four-six week courses of doxycycline, but this cannot be implemented in current mass drug administration programs. The purpose of this study is to evaluate if a shorter course (five days) with antibiotics that could be used in children and potentially pregnant women would likewise be effective.

Guatemalan patients with onchocercal nodules will be enrolled in an open label trial with four treatment groups: Group A (rifampin 20 mg/kg by mouth [po; maximum 600 mg/day]); B (azithromycin 12 mg/kg po [maximum 500 mg/day]); C (combination of rifampin 20 mg/kg po [maximum 600 mg/day] and azithromycin 12 mg/kg po [maximum 500 mg/day]); D (control group, multivitamin). At the end of the five day treatment course all participants will receive a single dose of ivermectin (150 mcg/kg).

Nodulectomies will be performed 9 months after treatment and the O. volvulus will be analyzed by immunohistochemical staining specific for Wolbachia.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant/non lactating females >5 years of age
* One onchocercal nodule in an anatomical position where it can be easily removed surgically

Exclusion Criteria:

* Pregnancy (based on urine pregnancy test)
* Breast-feeding
* Women taking oral contraceptives
* Allergy or other adverse reaction to either medication
* Use of other medications that might interact with rifampin
* Clinical evidence of liver disease (jaundice, swollen abdomen)
* Clinical evidence of chronic disease/alcoholism

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80
Dates: Start 2003-07; Study Completion 2004-05

PRIMARY OUTCOMES:
Eliminating Wolbachia endobacteria present in O. volvulus worms after 9 months

SECONDARY OUTCOMES:
Elimination of microfilaria in skin snips and histological examination of worms after 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Josef Amann, MD, MPH, Principal Investigator — CDC/NCID/DPD
Locations (1):
- Universidad del Valle/MERTU, Guatemala City, Guatemala